CLINICAL TRIAL: NCT07324590
Title: Thermal Imaging in the Diagnosis of Acute Testicular Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seinajoki Central Hospital (Other)
Collaborators: Hospital District of Helsinki and Uusimaa (Other); Turku University Hospital (Other Government); Kuopio University Hospital (Other); Oulu University Hospital (Other); Tampere University Hospital (Other); Pori Central Hospital (Unknown); Jyväskylä Central Hospital (Other)
Responsible Party: Principal Investigator, Mika Raitanen, Associate Professor, chief clinician, Seinajoki Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R25054L
Record Dates: First submitted 2025-11-21; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Testicular Diseases
Keywords: Testicular torsion; epididymites; testicular appendages torsion; Testicular pain
MeSH Terms: conditions — Testicular Diseases; Spermatic Cord Torsion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with acute testicular pain (Experimental)
  Interventions: Device: Thermidas thermal camera

INTERVENTIONS:
Device: Thermidas thermal camera — This kind of study has not been perfomed before

SUMMARY:
Acute scrotal pain due to testicular torsion is a rare but urgent urological condition that requires immediate surgery to prevent permanent damage or loss of the testicle. Early detection is crucial to minimize delays from the onset of pain to operative treatment. The diagnosis of torsion involves a combination of physical examination and imaging studies, such as Doppler ultrasound (DU). However, DU requires an experienced radiologist and may cause unnecessary time delays. Thermal imaging is a noninvasive technique that can detect skin surface temperature variations using a highly sensitive infrared camera. Although there are some promising animal studies using thermal imaging for the diagnosis of testicular ischemia, number of studies in humans is very limited.

According to a small pilot study in 2024, thermal imaging is a fast, feasible and noninvasive diagnostic tool that seems to have considerable potential in the evaluation of patients with acute testicular pain, especially those with symptoms of testicular torsion. However, further research with a larger sample size is needed. In this multicenter study, the investigators aim is to determine the role of thermal imaging in the diagnosis of acute testicular pain.

Males with acute testicular pain entering emergency are included. After informed consent thermal image of testicles will be taken before any additional investigations such as laboratory tests and DU. Participants are treated as usual and testicular temperatures will be correlated with final diagnosis after approximately 6-month study period is over.

DETAILED DESCRIPTION:
Acute testicular pain can have several causes, such as testicular torsion, but current diagnostic methods, such as DU, may be time-consuming and operator-dependent. The aim of this study is to evaluate the use of thermal imaging as a diagnostic tool for acute testicular pain, particularly in diagnosing testicular torsion, which requires urgent surgical treatment. Thermal imaging is a quick and non-invasive alternative that may help to reduce diagnostic delays. Results from two animal studies and a small pilot study conducted on patients in 2024 suggest that a thermal camera may be able to distinguish testicular torsion from epididymitis, which is another common cause for acute testicular pain. This multicenter study investigates the usability, accuracy, operator independence, and clinical applicability of thermal imaging in diagnosing acute testicular pain. According to a preliminary calculation, at least 146 participants are required with 80% statistical power and a 5% error rate. The sample size will be reassessed after six months, and if necessary, the enrollment phase will be extended.

A prospective 6-month study on the use and feasibility of thermal imaging for the diagnosing the cause of acute testicular pain will be conducted. Participating centers will include all university hospitals in Finland (Helsinki, Turku, Oulu, Tampere and Kuopio) and central hospitals of Seinäjoki, Jyväskylä and Pori. The study population will include all male participants presenting with acute testicular pain.

Participants with testicular pain are examined with thermal imaging immediately after arriving in the emergency department and before any other examinations (e.g., laboratory tests, DU). The results of the thermal imaging are not used in clinical decision-making; instead, they are compared later with the final diagnosis. Thermal imaging therefore does not influence the examinations or treatment decisions made for the participants, nor does it expose the participants to harmful ionizing radiation.

After entering the emergency room, the participants are verbally informed of the ongoing study and given research information sheet and preparatory instructions concerning the potential thermal imaging. The instructions explain how to tape the penis upward against the abdomen for 5 minutes to eliminate its thermal effect on the thermal image of the testicles. The trained and delegated research staff members give further verbal information about the study and the thermal imaging. Afterwards they collect the verbal permission and a signed informed consent form to take the thermal image. Participant's social security number, date, time and the code of the thermal image are written down on the consent form, which is stored in a secure place for safekeeping. Duplicate of the consent form remains with the participants. The estimated time needed for taking the thermal image is few minutes. Temperature results, however, will have no effect on decision making, as participants will be diagnosed and treated as usual using established routine diagnostic tools such as clinical evaluation, laboratory and urinary testing and DU.

A class IIa CE-approved Thermidas handheld camera (IRT-384 Tablet) will be used. It is designed for healthcare professionals to monitor and evaluate skin surface temperatures. The company Thermidas will educate our research staff in the use of their thermal camera. The leasing cost is 500 € per camera per month and it is covered by reaserch funf of Tampere University Hospital. The role of the company Thermidas in this study is to solely provide the thermal cameras for a fee, including the education in the use of the camera, and to store the images securely. The investigators have got a authorization for medicinal device from Fimea and approval from the ethics committee of Tampere University Hospital.

Technical specifications of the IRT-384 camera:

* Tablet operatin system: android
* Thermography sofware: Thermidas VistaClinic
* Display size: 10.1"
* Display resolution and colors: 1920 x 1200 pixels, 16 M colors
* RAM and ROM: 4 Gb and 64 Gb
* Connectivity: Wi-Fi
* Thermal camera resolution: 384 x 288 pixels
* Total active pixels: 110592
* Thermal Sensitivity(NETD: <0.05 C @ 30 C
* Accuracy: +- 2 C
* Field of View: 41.5 x 31.1
* Weight: 1.4 kg

The distance from the camera to the scrotum is approximately 20 cm while participant is standing, and testicles are hanging freely. Results of thermal imaging (temperature difference between testicles in Celsius) will be correlated with final diagnose at the end of study. Thermal picture (testicular temperatures) will be analyzed by two independent investigators blinded to each other and results will be correlated with the final diagnoses. SPSS statistical software will be used and sensitivity and specificity for thermal imaging will be calculated. Study registry holder will be Central Hospital of Seinäjoki.

Sub-study 1 Adult participants having funicular orchiectomy due to testicular cancer will be included. At operation thermal picture of untouched testicles will be taken before ligation or closure of the funicle (baseline) and at 5, 10 and 15 minutes afterwards. After this, funicular orchiectomy is performed as usual.

ELIGIBILITY:
Inclusion Criteria:

* Males, who come to emergency department due to acute testicular pain and sign informed consent.

Sub-study 1: Adult males, who are having funicular orchiectomy due to testicular cancer and sign informed consent.

Exclusion Criteria:

* Previous surgery or other operative procedure such as puncture in scrotal area within 30 days.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine role of thermal imaging in the diagnoses of acute testicular pain. To evaluate the effect of funicular ligation on testicular temperature (substudy 1). | Thermal picture is taken once at baseline. In substudy 1, thermal pictures of testicle will be taken at 0, 5, 10 and 15 minutes
  Temperatures of testicles
  * Comparison of temperatures (temperature diffrence) in Celsius of symptomatic and asymptomatic testicles
  * Temperatures of testicle in Celsius before and 5, 10 and 15 minutes after ligation of funicle (substudy 1)

CONTACTS AND LOCATIONS:
Overall Officials: Mika P Raitanen, M.D., Ph.D, associate prof, Study Chair — Seinöjoki Central Hospital
Locations (1):
- Hanneksenrinne 7, Seinäjoki, Finland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Background] Brooks JP, Brooks JM, Seals T. Smartphone Thermal Imaging in the Detection of Testicular Ischemia. Urology. 2021 Nov;157:233-238. doi: 10.1016/j.urology.2021.02.031. Epub 2021 Mar 6. PMID 33689763